CLINICAL TRIAL: NCT02851602
Title: Phospholipid and Sphingolipid Composition of High-density Lipoproteins (HDL) in Obese Non-diabetic Patients With Metabolic Syndrome
Acronym: SPHINGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VERGES 2013
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Blood Specimen Collection

ARMS (2):
- Obese (Experimental)
  Interventions: Biological: Blood sample
- control (Placebo Comparator)
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample

SUMMARY:
HDL in obese non-diabetic patients show major alterations in their function and thus their cardio-protective effects. These alterations could be explained by the quantitative and qualitative anomalies in the phospholipids and sphingolipids in the HDL. These molecules play a major role in HDL function and probably present early modifications in obesity, even before the onset of glycaemia deregulation.

The aim of this study is to show the presence of qualitative and quantitative modifications of phospholipids and sphingolipids in HDL from obese patients compared with HDL from non-obese controls.

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years
* fasting glycaemia < 1.10 g/l
* waist circumference > 102 cm for men and 88 cm for women (criteria NCEP/ATP III)
* 2 criteria among the following 3 (NCEP/ATP III criteria for metabolic syndrome):
* triglyceridaemia ≥ 1.50 g/l
* HDL cholesterol < 0.40 g/l for men and 0.50 g/l for women
* arterial blood pressure ≥ 130/85 mmHg or treatment for arterial hypertension
* patients who have provided written consent INCLUSION CRITERIA FOR HEALTHY SUBJECTS
* age > 18 years
* fasting glycaemia < 1.10 g/l
* waist circumference < 102 cm for men and 88 cm for women
* triglyceridaemia < 1.50 g/l
* HDL cholesterol ≥ 0.40 g/l for men and 0.50 g/l for women
* Healthy subjects who have provided written consent

Exclusion Criteria:

* Persons without national health insurance cover
* Diabetes
* Diseases that interfere with lipoprotein metabolism (dysthyroidism not controlled with the treatment, kidney or liver disease)
* Treatments that interfere with lipoprotein metabolism (lipid-lowering agents, oestrogens, corticoids, retinoids, antiretroviral agents)
* Pregnancy/breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Difference in the mass percentages of total phospholipids + sphingolipids compared with the total HDL mass | At inclusion
  in patients with abdominal obesity without hyperglycaemia compared with healthy controls

SECONDARY OUTCOMES:
Difference in the percentage of each family of phospholipids or sphingolipids compared with total phospholipids + sphingolipids | At inclusion
  in patients with abdominal obesity but without hyperglycaemia compared with healthy controls
Difference in the percentage of each sub-family according to the nature of the fatty acids for phosphatidylcholines on the one hand and sphingomyelins on the other in patients | At inclusion
  with abdominal obesity but without hyperglycaemia compared with healthy control

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France